CLINICAL TRIAL: NCT04875091
Title: Understanding Drivers of Variability in Treatment Response Among Emerging Adults in Behavioral Obesity Treatment
Brief Title: Understanding Variability in Behavioral Weight Loss Treatment Response in Young Women (Ready SET Health)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20018520
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Weight Loss; Weight Change, Body; Overweight or Obesity
Keywords: emerging adults; women; weight loss barriers
MeSH Terms: conditions — Weight Loss; Body Weight Changes; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Ready SET Health

INTERVENTIONS:
Behavioral: Ready SET Health — This behavioral weight loss intervention will span 16 weeks. The first session (Week 1) will be a virtual "Weight Loss 101" group kick-off followed by 15 weeks of a technology-mediated program consisting of the following: weekly emailed content (videos and readings explaining key skills and strategies to produce weight loss) and weekly emailed tailored feedback (based on self-monitoring data from participants). A trained interventionist ("coach") will lead the group session, provide weekly tailored feedback, and monitor participant progress.

SUMMARY:
This study is a single-arm behavioral weight loss intervention for emerging adult women with in-person assessments at 0 (baseline) and 4 months (post-treatment) in addition to EMA data collection regarding risk factors known to interfere with program engagement and weight loss in this high-risk population (e.g., sleep, psychological distress, life events).

DETAILED DESCRIPTION:
This study will implement a 4-month Internet-based behavioral weight loss intervention in order to collect ecological momentary assessment (EMA) data that will shed light on real-time barriers to weight management. The intervention is evidence-based and adapted with respect to content and delivery mode in order to meet the needs of emerging adult women. Consenting and eligible participants will receive 1 virtual group session led by a trained interventionist followed by weekly emails directing them to an intervention website housing video and .pdf content, weekly text messages, emailed tailored feedback regarding their weight loss behaviors and progress, and a closed Facebook group to facilitate social support. All participants will be followed for 4 months with hybrid in-person/virtual assessments at 0 and 4 months; in addition, all participants will be asked to respond to EMA prompts throughout the 4-month intervention period (Week 2, Week 4, Week 7, and Week 13).

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years of age
* BMI (body mass index) 25-45 kg/m2
* Female gender identity

Exclusion Criteria:

* Report of uncontrolled medical condition that may pose a safety issue given the recommendations for the diet and unsupervised physical activity
* Diagnosed cardiovascular or metabolic disease
* Report of a heart condition, chest pain during periods of activity or rest, or loss of consciousness
* Recent change in use of medications that may impact weight or metabolic function
* Cancer in the past 5 years, except non-melanoma skin cancers or early-stage cervical cancer
* Current symptoms of alcohol or other substance dependence
* Report of diagnosis or history of Anorexia Nervosa or Bulimia Nervosa, or any compensatory behaviors within the previous 3 months
* Hospitalization for depression or other psychiatric disorder within the past 12 months
* Lifetime history of bipolar disorder or psychotic disorder
* Planning to move from the area within the study period
* Currently pregnant, pregnant within the past 6 months, currently breastfeeding or planning to become pregnant within the next 6 months
* Current involvement in a weight loss program or current use of weight loss medication
* Recent significant weight loss
* Inability to read or speak English
* Lack of a smartphone or unwillingness to use it for study components

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female gender identity
Enrollment: 48 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Weight change | 4-months (post-intervention)
  Percent weight change (fasting weight in kg, measured in-person by trained assessors)

SECONDARY OUTCOMES:
Weekly weight change | 4-months (throughout intervention)
  Weekly weight change (weight in lbs obtained through participants' Bluetooth-/wireless-connected study scale; converted to kg for analyses)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No